CLINICAL TRIAL: NCT05109273
Title: Atrioventricular Nodal Reentrant Tachycardia Ablation With irrigATEd catheteR And Three-dimensional elecTroAnatomiC Mapping (WATER ATTAC)
Brief Title: Atrioventricular Nodal Reentrant Tachycardia Ablation With Irrigated Catheter and Three-dimensional Electroanatomic Mapping
Acronym: WATER ATTAC
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Bertini, Principal Investigator, University Hospital of Ferrara
Other Study IDs: 676/2021/Oss/AOUFe
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Atrioventricular Nodal Re Entrant Tachycardia
Keywords: AVNRT; Ablation; Electroanatomical mapping system; Irrigated catheter; Radiofrequency; Arrhythmias; Electrophysiology; SVT; Slow-Fast
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transcatheter ablation — Three-dimensional electroanatomic mapping and radiofrequency ablation with irrigated catheter

SUMMARY:
The WATER ATTAC study aims at multicentric, longitudinal, perspective evaluation of safety and efficacy of atrioventricular nodal reentrant tachycardia (AVNRT) performed combining irrigated ablation catheter and three-dimensional electroanatomic mapping system. Efficacy and rate of complications will be evaluated over medium and long term follow-up.

DETAILED DESCRIPTION:
Atrioventricular nodal reentrant tachycardia (AVNRT) is the most common supraventricular tachycardia in clinical practice, more common in women than in men. It can occur at all ages, but it is more likely to begin in young adults, with average age of onset around 32 years. Due to its sudden onset and cessation it is classified in the group of paroxysmal supraventricular tachycardias (PSVT), accounting for almost two thirds of the total.

AVNRT is a regular supraventricular tachycardia resulting from formation of reentry circuit confined to atrioventricular node and perinodal atrial tissue. About 80-90% of patients with AVNRT have the common form of arrhythmia, also called "typical" or "slow-fast" type.

Slow-fast AVNRT usually begins when premature atrial complex (PAC) arrives at AV node when fast pathway is in its refractory period. Therefore, antegrade conduction along fast pathway is blocked. If premature beat arrives in specific time window, slow pathway, with shorter refractory period, is available for conduction to ventricle. Premature beat leads through slow way, and, through final common way, to His bundle. As a result, PR interval of premature beat will be longer than normal beats conducted through fast track. If fast pathway has recovered its excitability by the time impulse of the slow pathway reaches distal junction of the two paths, impulse can lead retrograde through fast pathway. Circuit can then become repetitive with antegrade conduction along slow pathway and retrograde conduction along fast pathway with consequent triggering of sustained tachycardia. This proposed mechanism explains series of clinical observations of AVNRTs: single PAC can initiate arrhythmia and in the same way penetration in reentry circuit by PAC can abruptly interrupt arrhythmia.

Up to 20% of patients with AVNRT have uncommon forms of arrhythmia, referred to as "atypical" AVNRT. There are cases in which antegrade conduction can occur along fast pathway with retrograde conduction along slow pathway (fast-slow type).

Some patients, on the other hand, have more slow pathways, in which both antegrade and retrograde pathways of circuit use slow AV nodal pathways (slow-slow type).

For patients with AVNRT episodes that occur frequently and are poorly tolerated or require hospitalization, the only chronic therapy recommended in class I by international guidelines is catheter ablation. Evidence from randomized trials has shown that catheter ablation is significantly superior to antiarrhythmic drug therapy in preventing hospital admission for recurrences of tachycardia at 5 years.

AVNRT catheter ablation is a procedure that involves cardiac mapping and subsequent ablation of the arrhythmic substrate. Cardiac mapping refers to the careful movement of a mapping or ablation catheter in the area of interest, probing site where ablation will be able to cure arrhythmia. Cardiac mapping during electrophysiological testing identifies temporal and spatial distributions of electrical potentials generated by myocardium during normal and abnormal rhythms. This process allows to describe spread of activation from its inception to its completion within a region of interest and, in its usual application, is focused towards identifying site of origin or critical site of conduction for arrhythmia. The recurrence rate after radiofrequency catheter ablation varies from 3.5 to 5.2% during a 6 - 24 months follow-up.

The most worrying complication related to AVNRT ablation is iatrogenic disturbance of atrioventricular conduction requiring pacemaker implantation. According to large recent trial, 3% of patients treated with AVNRT ablation underwent pacemaker implantation during a median follow-up of 4 years [9]. In particular, the risk of pacemaker implantation is present not only in the periprocedural period, but persists during the long-term follow-up.

Since the first description of radiofrequency ablation directed to site of slow pathway and guided by fluoroscopic anatomical landmarks or intracardiac electrograms, technique for AVNRT ablation has been implemented in years. One of the major improvements was three-dimensional electroanatomic mapping. Electroanatomic (or electromagnetic) mapping, available in many electrophysiology laboratories, is based on use of special catheter with locatable sensor tip, connected to mapping and navigation system. The system can generate color-coded static maps or animated dynamic maps of activation wavefront. These images can define reentrant circuits as well as site of origin of ectopic activity with centrifugal, regional or asymmetric diffusion of electrical activity. A major advantage of three-dimensional electroanatomic mapping is its ability to allow catheter to anatomically and accurately "revisit" critically important recording site previously identified during electrophysiological study, even if tachycardia is no longer present or inducible. This accurate repositioning can allow further application of the radiofrequency current to critical sites that otherwise cannot be performed with high degree of accuracy and reproducibility. Furthermore, direct visualization of anatomical structures such as coronary sinus ostium, tricuspid anulus and bundle of His allows to delineate in precise and 3D way the Koch triangle, which is crucial a reference to perform ablation of slow pathway without affecting the atrioventricular node.

Three-dimensional electroanatomic mapping system also reduces or avoids radiation exposure and improve accuracy in localization and ablation of target site by means of three-dimensional visualization of anatomical map, with high success rates and reducing rate of complications and recurrences. The use of three-dimensional electroanatomic mapping has been associated with significant reduction in patient radiation dose, operator radiation dose, and total fluoroscopy time.

Another technical improvement was irrigation of distal electrode of ablation catheter with saline and heparin, which reduced the risk of complications such as thrombus and steam pop formation. While in non-irrigated catheters, energy delivery is limited by temperature at catheter-tissue interface, irrigated catheters allow for greater energy delivery and create deeper lesions. Use of irrigated catheters for AVNRT ablation increased from 0% in 2005 to 23% in 2015 but still remains low. Combination of irrigation and flexible tip allows stable contact with myocardial tissue with uniform delivery of radiofrequency and continuous cooling.

In 2019, our group released an initial report on efficacy and safety of AVNRT ablation with new flexible tip open irrigated catheter (FlexAbilityTM, Abbott, St. Paul, MN, USA) combined with 3D EAM system (EnSite PrecisionTM, Abbott, St. Paul, MN, USA).

Our study demonstrated the efficacy and safety of flexible tip open irrigated catheter ablative technique used in combination with 3D EAM. Our group recently published a subsequent work on a larger cohort of patients with long-term follow-up. About 150 patients were enrolled with mean follow-up period of 38 months. Acute procedural success rate was 96.7% (145/150 patients). During follow-up, 11 patients experienced arrhythmia recurrence (7.3%). No patient developed atrioventricular conduction block requiring pacemaker implantation (0%). In our study, therefore, results related to acute procedural success and long-term follow-up showed that AVNRT can be treated safely and effectively with irrigated flexible tip catheters and 3D EAM.

With the WATER ATTAC study we want to verify if the same results can be obtained by expanding the sample size in a multicentric context, with the aim of externally validating AVNRT tranascatheter ablation procedure with irrigated catheter and three-dimensional electroanatomic mapping.

The purpose of this study is to prospectively evaluate safety and efficacy of AVNRT ablations performed by combining irrigated catheter with three-dimensional electroanatomic mapping system. The effectiveness of procedure and incidence of complications in medium and long term follow-up will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing electrophysiologic study (EPS) for paroxysmal supraventricular tachycardia
* evidence of dual AV node pathway or atrioventricular nodal reentrant tachycardia (AVNRT) induction at EPS
* Attempt of AVNRT ablation with irrigated catheter and three-dimensionale electroanatomic mapping system

Exclusion Criteria:

* Age <18 years
* Ablation with non-irrigated catheter
* Ablation without electroanatomic mapping system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing EPS for SVT, with confirm of AVNRT at EPS, treated with transcatheter ablation by means of irrigated catheter and 3D electroanatomic mapping system
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 12 months
  Recurrence of AVNRT during follow-up
Procedural complication | 12 months
  AV iatrogenic block

SECONDARY OUTCOMES:
Acute success rate | Immediate post-procedure
  Non-inducibility of AVNRT or absence of dual AV node pathway

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertini, MD, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, Italy